CLINICAL TRIAL: NCT00713570
Title: the Cognitive Ability Dose Associate With COMT, 5HT6, BDNF and Biological Systemic Pathway Candidate Genes in General Population
Brief Title: Explore the Nature Factors Relevant to Learning-Pioneering Natural Factors That Influences Science Learning II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital Research Ethics Committee, National Taiwan University Hospital
Other Study IDs: 200612069R
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: intellectual functioning; memory,visual-spatial and perceptual functions; cognitive abilities; COMT; BDNF; neuron biological systemic pathway candidate genes; Chinese; Taiwan; Healthy subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A,1,II

SUMMARY:
Genetic research has provided the most exciting breakthroughs in neuroscience and cognitive science. Partially genetically determined cognitive impairments have been described in people with COMT, 5HT6, BDNF (Swillen et al., 2000; Moss et al., 1999, Henry et al., 2002, Bilder et al., 2002)and biological systemic pathway candidate genes.

Selective inhibitors of COMT proved to improve cognitive function in animals and in patients with Parkinson's disease (Carlsson, et al, 2000). Recent studies suggested that variation in COMT activity might have neurobiological effects specific to the prefrontal cortex; the COMT (Val) allele with high activity impairs tasks of prefrontal cognition in people with schizophrenia (Egan et al., 2001) and higher loading of the COMT (Met) allele is associated with better cognitive performance on attention and processing speed in people with chronic schizophrenia (Bilder et al., 2002). Moreover, prefrontal dopamine levels are increased in COMT knockout mouse model (Gogos et al., 1998). This suggests that in people who have heterozygosis on COMT, dopamine levels could be abnormal. Thus, variation in COMT expression could also affect performance on prefrontal cognitive tasks. In the previous study, we found the neuropsychological profile in students with COMT (Met) allele is better in object perception, problem solving and planning, and abstract and social thinking (Henry et al., 2002).

5-HT6 inhibitor has been reported to raise extracellular acetylcholine levels in the cortex and hippocampus (Dawson et al., 2001 and Riemer et al., 2003). Acetylcholine release in hippocampal and cortical regions is known to be important for memory acquisition and retention, and several groups have demonstrated that 5-HT6 blockade overcomes scopolamine-induced amnesia. We hypothesize that variations in COMT and 5-HT6 are associated with genotype that will cause a poor/better performance in cognitive tasks.

With the aim to establish the possible correlation between candidate genes (COMT, 5HT6,BDNF and biological systemic pathway candidate genes. etc) and cognitive ability, which will provide us an understanding on factors and its extent that affect students' thinking, and then develop appropriate teaching models or strategies for assisting students in learning. It seems timely, therefore, to consider how we might implement our increased understanding of brain development and brain function to explore educational questions.

DETAILED DESCRIPTION:
In the past decade, the number of studies concerning the connections between neuroscience and cognitive science has been growing dramatically. The findings might inform us how learners find a better way to learn. However, it has been proven that it is difficult to apply these findings to the real classrooms (Bruer, 1997; Goswami, 2006). This is mainly because learning behavior requires interactions among various cognitive abilities, yet most neuroscience-related research stressed only on a cognitive ability or microstructure alone. In other words, neuroscience research often focuses on microstructure of cells, while cognitive research focuses on systematic integrations. Generally speaking, a single-neuron cell is insufficient for behavior development.

Based on the statement, "whole does not equal to sum of every single part", simply examining a microstructure will not lead to an understanding of behavior that produced by cell assembly/synergy. The current neuroscience technology for detecting activities in two or more cells simultaneously is still in progress, and issues on how cells can work harmoniously have been seriously considered recently. Clearly, educators do not study learning at the level of the cell. A successful learning depends on the curriculum, the teacher, context provided by the classroom and the family, and the context of the school and the wider community. All of these factors synergistically interact with the characteristics of individual brains. For example, children with high levels of the monoamine oxidise A who experience maltreatment and adverse family environments seemed to be protected from developing antisocial behavior (Caspi, et al., 2002), possibly via moderating effects on their neural response to stress. Diet is also reported to affect the brain. A child whose diet is poor will not be able to respond to excellent teaching in the same way as a child whose brain is well-nourished. It is already possible to study the effects of various medications on cognitive function. Methylphenidate (Ritalin) has been shown to improve stimulus recognition in children with ADHD (Attention Deficit Hyperactivity Disorder) (Seifert, et al., 2003). Neuroimaging techniques also offer the potential to study the effects of different diets, food additives and potential toxins on educational performance. In our opinion, applying neuroscience findings to actual classroom will be beneficial to students in learning. It will be of value if studies about the connections between neuroscience and education can be extended to other related topics, such as practical mechanisms, which will result in a meaningful integration. Therefore, exploring the behavior-cognitive-neuron-gene system (BCNG system) (Fig 1) and developing science educational theories from neuroscience-related studies will be the main objectives and long-term goads as a result of our future research.

The BCNG system includes two main categories, namely "science education" and "neuroscience". Currently, science education research including our previous endeavors emphasizes how cognitive abilities affects learners' academic achievement and performance (for example, Wang, Chang, & Li, published online; Chang et. al., 2006) while neuroscience stresses on the relationships between individual's cognitive ability and neurophysiology/ biochemistry mechanism. Currently, there are ten aspects about cognitive ability, including intelligence, attention, memory, linguistic ability, spatial ordering, higher order cognition, ordering system, action system, social interaction system and emotion. These aspects can be divided further into sub-topics.

Changes on cognitive ability are caused both by innate, genetic inherence of learning ability and acquired ability enforced by learning. However, researchers have not yet clearly understood the extent that innate and acquired factors influence an individual's cognitive abilities.

In learning process, students who do not perform well in academic as other students due to poor cognitive ability will affect their willingness to learn. In other words, low cognitive ability will affect students' willingness to learn. Deficiencies in linguistic system( includes defects in listening, speaking, reading and writing), elements that affect language skills (containing disabilities in phonemes, morphemes and syntax), and disagreements in activities of muscles (which cause messy in writing) will make students considered to be clumsy and indolent or teased by peers and lead to decreased learning motivation. Therefore, Livan(2001) asserts that educationists should first understand each student's innate cognitive ability, and then give a priority to develop a subject that matches a student's cognitive ability, so that a student's learning interest and achievement outcome will be raised, and eventually this model/strategy will also work for the subjects that do not actually match student's cognitive ability. This suggestion is, to some extent, in alignment with our previous work (Chang and Tsai, 2005), which we found that teacher-centered instructional approach seemed to enhance more positive attitudes of less constructivist-oriented learning preferences students, whereas the student-centered method was more beneficial to more constructivist-oriented learning preferences students on their attitudes toward earth science in a computer-assisted learning environment. In the process of developing and undertaking the BCNG system, this research project starts with innate factors that might affect learners' cognitive ability. Based on the understanding of relationships existed between cognitive ability and genotypes of possible cognition-related genes, appropriate instructional models or strategies might be appropriately developed to better assist/match students' learning.

1. Using existing test batteries to understand subjects' intellectual functioning, memory,visual-spatial and perceptual function, executivefunction, attention and science problem-solving ability.
2. Identifying genetic polymorphism of human COMT, BDNF, 5-HT6 and other genes in Taiwan by investigating single nucleotide polymorphism (SNPs) of the genes among Taiwanese subjects using PCR and DNA sequencing.
3. Screening and comparing the allelic distribution of each SNP among tested subjects and exploring if there is cognitive-associated SNP(s) in these gene.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with inform concern

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Taiwan genernal population
Sampling Method: Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2006-08; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
observational studies, related to core objectives of the study and learning. | at least five years follow

CONTACTS AND LOCATIONS:
Overall Officials: Chung Yi Hu, PhD, Principal Investigator — Department of Clinical Laboratory Sciences and Medical Biotechonology; Chun-Yen Chang, PhD, Principal Investigator — Professor of Department of Earth Sciences Director of Science Education Center,PI of Building the e-Learning Research Teams for Excellence National Taiwan Normal University; Ting-Chi Yeh, MD, Principal Investigator — Division of Pediatric Hematology-Oncology, Mackay Memorial Hospital
Locations (1):
- Chung-Yi Hu, Taipei, Taiwan